CLINICAL TRIAL: NCT03054727
Title: Long Term Natural History of PTS and Other Adverse Outcomes After Venous Thromboembolism in the Optimev Study (SPOT)
Brief Title: Long Term Assessment of Post Thrombotic Syndrome : OPTIMEV Study ( SPOT )
Acronym: SPOT
Status: Completed | Type: Observational
Sponsor: Association des Médecins Vasculaires Hospitaliers (Other)
Collaborators: Daiichi Sankyo (Industry); Ministry of Health, France (Other Government); LEO Pharma (Industry); Sanofi (Industry); University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: OPTIMEV SPOT
Record Dates: First submitted 2016-09-20; First posted 2017-02-16 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Post Thrombotic Syndrome; Venous Thromboembolism; Cardiovascular Diseases
Keywords: Post Thrombotic Syndrome; Venous Thromboembolism; Incidence; Risk factors; Venous ulcer
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thromboembolism; Cardiovascular Diseases; Varicose Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Villalta phone score > or = to 5: patients with VTE in the OPTIMEV cohort with an Utne and Sandset Villalta phone score > or = to 5 at the end of the follow-up call AND a random selection of patients free from any VTE after the first 3 years of follow-up in OPTIMEV with an Utne and Sandset Villalta phone score > or = to 5 at the end of the follow-up call
  Interventions: Other: Villalta phone score > or = to 5; Other: Villalta phone score < 5
- Villalta phone score < 5: patients with VTE in the OPTIMEV cohort with an Utne and Sandset Villalta phone score < 5 at the end of the follow-up call AND random selection of patients free from any VTE after the first 3 years of follow-up in OPTIMEV with an Utne and Sandset Villalta phone score < 5 at the end of the follow-up call
  Interventions: Other: Villalta phone score > or = to 5; Other: Villalta phone score < 5

INTERVENTIONS:
Other: Villalta phone score > or = to 5 — Follow up call. At the end of the follow-up, the patients who received an Utne and Sandset Villalta phone score > or = 5 will have a visit with clinical and CUS assessments of PTS/ venous insufficiency.
  All patients will have self administered-questionnaires. For Grenoble Center, the 200 first patients with clinical follow-up will have an Echo-Doppler examination.
  Other Names: Clinical Follow-Up Group
Other: Villalta phone score < 5 — Follow up call. At the end of the follow-up, the patients who received an Utne and Sandset Villalta phone score < 5, will don't have a clinical follow up.
  All patients will have self administered-questionnaires.
  Other Names: No Clinical Follow-Up Group

SUMMARY:
Post-thrombotic syndrome (PTS) is a frequent and burdensome complication of deep-vein thrombosis (DVT). In the absence of curative treatment of established PTS, its management is based on the prevention of its occurrence thanks to anticoagulants and compression stockings.

So far, predictors of disabling PTS are unknown precluding from optimally selecting patients for invasive (early thrombus removal) or innovative/expensive treatments. In addition, little is known on the incidence of PTS in the very long-term.

Objectives: To assess, 12 years after a symptomatic venous thromboembolic (VTE) event, Primary objective: incidence and severity of PTS after a lower limb DVT.

Main Secondary objectives:

1. Incidence and severity of PTS according to VTE initial presentation (isolated distal DVT, isolated proximal DVT, PE + DVT).
2. Incidence and risk factors of disabling PTS Methods: Very long-term follow-up (12 years) of patients recruited in the large, multicentre, prospective, observational OPTIMEV study for a suspicion of VTE confirmed or ruled out with objective tests (Clinical Trials NCT00670540).

All patients with a DVT, an isolated PE and a random selection of controls (VTE - patients without any history of VTE after the 3 years of follow-up) will first benefit from a phone-PTS assessment. Those patients presenting at least a mild venous insufficiency and a selection of controls will undergo a clinical follow-up visit with clinical and Compleat Ultra Sound (CUS) assessment of PTS/venous insufficiency and an assessment of quality of life.

Perspectives: Improving our knowledge of PTS' incidence and predictors and of the impact of usual treatment. Better selecting patients eligible for invasive/innovative/expensive preventative procedures.

DETAILED DESCRIPTION:
Post thrombotic syndrome (PTS) refers to chronic manifestations of venous insufficiency following a deep vein thrombosis (DVT). It is the most frequent complication of DVT, which affects up to 40% of patients after a proximal DVT (popliteal veins and above).

Though not lethal, PTS is burdensome and severly impacts patient's quality of life (QOL). In addition after a DVT, PTS was found to be an important predictor of total and medical costs. Thus PTS is not just a cosmetic problem and constitutes a real public health concern in the field of VTE. However, so far, many epidemiologic and therapeutic issues remain unresolved.

On an epidemiologic point of view, incidence of PTS in the long term (i.e. after 5 years) is largely unknown. In addition, there is no available reliable data on the risk of PTS after isolated distal DVT (i.e. infrapopliteal DVT without pulmonary embolism (PE), >50% of all lower limb DVT) or isolated PE. At last, risk and independent predictors of the most severe disabling forms of PTS (particularly venous claudication and venous ulcers) need to be assessed (absence or old and outdated data).

On a therapeutic point of view, so far there is no curative treatment of established PTS. The cornerstone of PTS' treatment lies on its prevention via an optimal anticoagulation therapy, the use of compression stockings (the effectiveness of which was recently questioned by the SOX RCT trial) and sometimes thrombolysis for cases of very proximal DVT without bleeding risk. Impact in the very long term of usual DVT treatment on PTS natural history, prescribed in routine clinical practice in a real life setting, has never been assessed. Furthermore, absence of identified independent predictors of disabling PTS constitutes an important break to the use and to assess the full effectiveness of invasive therapies.

In this perspective, the investigators aim performing a very long term follow-up (12 years) of the already constituted OPTIMEV cohort in order to try to answer most of the above-mentioned epidemiologic and therapeutic unresolved issues.

Objectives Primary objective: To assess incidence (from baseline till up to 12 years) and severity of PTS, 12 years after a lower limb DVT, calculated with the clinical Villalta score.

Secondary objectives: To assess in the very long term (12 years)

1. Determine risk factors of disabling PTS (DVT patients).
2. Characterize the incidence and severity of PTS according to VTE initial presentation (isolated distal DVT, isolated proximal DVT, PE + DVT).
3. Determine the rate of venous insufficiency in the unexposed population and also in the exposed population.
4. Estimate the impact of PTS on patient's quality of life.
5. Assess the incidence of cancers in the population, by comparing exposed patients and non exposed patients included in OPTIMEV cohort.
6. Assess the incidence of cardiovascular events in the population, by comparing exposed patients and non exposed patients included in OPTIMEV cohort.
7. Assess the incidence of death in the population, by comparing exposed patients and non exposed patients included in OPTIMEV cohort.
8. Assess the incidence of new DVT in the population, by comparing exposed patients and non exposed patients included in OPTIMEV cohort.
9. Assess the attributable risk of DVT to the signs and symptoms of chronic venous insufficiency in DVT patients
10. Determine whether there is a correlation between CUS findings and PTS clinical severity in 200 patients with PTS (Villalta > or = 5).
11. Measure the incidence of hemorrhage events in the population, with comparison between exposed and non exposed patients included in OPTIMEV cohort.

Methods Cohort study of exposed and unexposed patients nested in the OPTIMEV multicentre observational study (Clinical Trials NCT00670540) Constitution of the OPTIMEV cohort: From November 2004 to January 2006, 8256 patients with a suspicion of symptomatic VTE (lower and upper extremity DVT, PE) were enrolled and benefited from objective tests to confirm or rule out the suspicion of VTE. This included a bilateral whole leg compression CUS for all cases of suspicion of DVT; Baseline characteristics including patient's demographics, signs, symptoms & risk factors for VTE, venous status, results of objective tests and treatments were prospectively collected in an electronic case report form.

Patients with a confirmed VTE and a random selection of controls (patients for whom VTE was ruled out at baseline) were initially followed up by phone by clinical research assistants during 3 years using standardized questionnaires to obtain information on health-related events (death, VTE recurrence, bleeding, arterial cardiovascular events, diagnosis of cancer or of lower limb ulcer, hospitalization and treatments). The general practitioner or the vascular medicine physician was contacted whenever a possible event was reported or when the patient's history seemed potentially unreliable. Medical records were reviewed in case of hospitalization or a new visit to the vascular physician during the follow- up period. All suspected adverse events were adjudicated by the study's expert committee.

At 3 years our rate of lost to follow-up or of patients who declined to continue the study was low (<3%) For this very long-term follow-up (12 years), patients with VTE and a random selection of patients free from any VTE will be considered.

As per previous follow-up visits, clinical research assistants will contact all eligible patients using the same standardized questionnaires and will assess PTS/venous insufficiency using a validated phone-questionnaire (Villalta score of Utne and Sandset). Patients with a suspicion of disabling PTS/venous insufficiency and a random selection of controls will be referred to a participating vascular medicine physician for a clinical follow-up visit with realization of a PTS assessment (Villalta score and CEAP) and a whole limb CUS exploration of the venous system + Ankle Brachial Index (ABI) measurement). QOL questionnaires will also be filled.

Statistical considerations Statistical analyses will be performed by the Themas team in Grenoble. Based on the results of a pilot-feasibility study (random selection of 100 VTE patients, 15% lost to Follow-Up (FU) and 5% of death), 1000 patients with lower limb DVT or PE at baseline ("exposed" patients) should attend the clinical follow-up visit. This will allow us to estimate, with a precision of plus or menus 3% an incidence of PTS at 12 years of 45% and with a precision of plus or menus 2.5% an incidence of disabling PTS of 20%.

Perspectives This study should improve our knowledge on the long term incidence of PTS according to various presentations of VTE disease, on the impact of routine clinical practice therapeutic management (particularly compression therapies and anticoagulation) on the risk of PTS, and should allow determining independent predictors of disabling PTS. On a clinical practice point of view, this study should assess the benefit of PTS preventative treatment after an isolated DVT or an isolated PE and to better selecting patients eligible for invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Exposed patients: Patients with a lower limb DVT and/or a PE
* Unexposed patients: Random selection of controls (1:1) free from any VTE event at the 3 years follow-up visit

Exclusion Criteria:

* Severe venous insufficiency at baseline (CEAP C5-C6)
* Severe lower limb peripheral arterial disease (critical limb ischemia)
* Altered mental status
* Decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study of exposed and unexposed patients nested in the propsective OPTIMEV cohort
Sampling Method: Probability Sample
Enrollment: 2475 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
disabling PTS | 12 years
  Clinical Villalta score > or = 10 (moderate or severe PTS) and/or venous claudication (Villalta score assessed during the clinical Follow-Up visit by a vascular medicine physician (signs) and by the patient (symptoms)

SECONDARY OUTCOMES:
Risk factors of disabling PTS | at inclusion
  Risk factors could be evaluated by the data base and the 3 years follow-up of the OPTIMEV cohort and with the follow-up call on medical history of the patient.
PTS severity | at inclusion
  PTS severity will be assessed with the Villalta scale :
  0-4 : no PTS ; 5-9 : mild PTS 10-14 : moderate PTS
  > or = to 15 or presence of ulcer: severe PTS
Incidence of venous insufficiency | at inclusion
  incidence of venous insufficiency will be evaluated with the CEAP classification and the analyse of collected signs and symptoms by the Utne and Sandset Villalta phone score.
Global Quality of life | at inclusion
  EUROQUOL questionnaire (generic questionnaire)
Specific Quality of life | at inclusion
  chronic venous disease quality-of-life (CIVIQ) questionnaire
Incidence of cancers | at inclusion
  number of cancers in the population. Information on cancer occurence will be collected during the phone follow-up
Incidence of cardio-vascular events (stroke, myocardial infarction, peripheral arterial disease) | at inclusion
  Description with the same definition of the 3-year-follow-up of OPTIMEV. The events will be adjudicated by the study expert committee composed of at the last two doctors, on the basis of medical reports
Incidence of deaths | at inclusion
  number of deaths in the population. Deaths data will be collected during the phone follow-up visit
Incidence of new thromboembolic disease | at inclusion
  The event will be adjudicated by the study expert committee composed of at the last two doctors, on the basis of medical reports
Attributable risk of DVT in PTS severity | at inclusion
  Assessed via the Villalta score by comparing exposed patients and non-exposed patients.
Doppler Ultrasound and PTS severity | at inclusion
  correlation between Doppler Ultrasound results (deep and/or superficial reflux , lack of recanalization or partial recanalization, parietal sequelae) and different levels of severity of PTS (mild , moderate and severe +/- venous claudication)
Incidence of hemorrhage events | at inclusion
  The event will be adjudicated by the study expert committee composed of at the last two doctors, on the basis of medical reports

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc JB Bosson, MD, PhD, Study Chair — University Hospital, Grenoble; Jean-Philippe JP Galanaud, MD, PhD, Principal Investigator — Montpellier University Hospital; Gilles GP Pernod, MD, PhD, Principal Investigator — University Hospital, Grenoble; Marie-Antoinette MS Sevestre, MD, PhD, Principal Investigator — Amiens University Hospital
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galanaud JP, Sevestre MA, Genty C, Pernod G, Quere I, Bosson JL. Is it useful to also image the asymptomatic leg in patients with suspected deep vein thrombosis?: comment. J Thromb Haemost. 2015 Nov;13(11):2127-30. doi: 10.1111/jth.13123. Epub 2015 Sep 30. No abstract available. PMID 26332772
- [Background] Galanaud JP, Arnoult AC, Sevestre MA, Genty C, Bonaldi M, Guyard A, Giordana P, Pichot O, Colonna M, Quere I, Bosson JL; OPTIMEV-SFMV Investigators. Impact of anatomical location of lower limb venous thrombus on the risk of subsequent cancer. Thromb Haemost. 2014 Dec;112(6):1129-36. doi: 10.1160/TH14-04-0351. Epub 2014 Aug 7. PMID 25104514
- [Background] Le Moigne E, Genty C, Meunier J, Arnoult AC, Righini M, Bressollette L, Bosson JL, Le Gal G; OPTIMEV Investigators. Validation of the LEFt score, a newly proposed diagnostic tool for deep vein thrombosis in pregnant women. Thromb Res. 2014 Sep;134(3):664-7. doi: 10.1016/j.thromres.2014.07.009. Epub 2014 Jul 17. PMID 25087889
- [Background] Galanaud JP, Sevestre MA, Genty C, Kahn SR, Pernod G, Rolland C, Diard A, Dupas S, Jurus C, Diamand JM, Quere I, Bosson JL; OPTIMEV-SFMV investigators. Incidence and predictors of venous thromboembolism recurrence after a first isolated distal deep vein thrombosis. J Thromb Haemost. 2014 Apr;12(4):436-43. doi: 10.1111/jth.12512. PMID 24450376
- [Background] Galanaud JP, Bosson JL, Genty C, Presles E, Cucherat M, Sevestre MA, Quere I, Decousus H, Leizorovicz A. Superficial vein thrombosis and recurrent venous thromboembolism: a pooled analysis of two observational studies. J Thromb Haemost. 2012 Jun;10(6):1004-11. doi: 10.1111/j.1538-7836.2012.04704.x. PMID 22429908
- [Background] Maufus M, Bosson JL, Genty C, Delluc A, Imbert P, Gagne P, Rolland C, Bressollette L, Le Gal G. [Validation of a deep vein thrombosis prediction rule in primary care]. J Mal Vasc. 2012 Feb;37(1):9-14. doi: 10.1016/j.jmv.2011.10.005. Epub 2011 Dec 12. French. PMID 22169238
- [Background] Galanaud JP, Genty C, Sevestre MA, Brisot D, Lausecker M, Gillet JL, Rolland C, Righini M, Leftheriotis G, Bosson JL, Quere I; OPTIMEV SFMV investigators. Predictive factors for concurrent deep-vein thrombosis and symptomatic venous thromboembolic recurrence in case of superficial venous thrombosis. The OPTIMEV study. Thromb Haemost. 2011 Jan;105(1):31-9. doi: 10.1160/TH10-06-0406. Epub 2010 Sep 30. PMID 20886192
- [Background] Utne KK, Ghanima W, Foyn S, Kahn S, Sandset PM, Wik HS. Development and validation of a tool for patient reporting of symptoms and signs of the post-thrombotic syndrome. Thromb Haemost. 2016 Jan;115(2):361-367. doi: 10.1160/th15-04-0318. Epub 2015 Sep 17. PMID 26422814
- [Background] Johnson SA, Stevens SM, Woller SC, Lake E, Donadini M, Cheng J, Labarere J, Douketis JD. Risk of deep vein thrombosis following a single negative whole-leg compression ultrasound: a systematic review and meta-analysis. JAMA. 2010 Feb 3;303(5):438-45. doi: 10.1001/jama.2010.43. PMID 20124539
- [Background] Galanaud JP, Sevestre MA, Genty C, Laroche JP, Zizka V, Quere I, Bosson JL; OPTIMEV SFMV investigators. Comparison of the clinical history of symptomatic isolated muscular calf vein thrombosis versus deep calf vein thrombosis. J Vasc Surg. 2010 Oct;52(4):932-8, 938.e1-2. doi: 10.1016/j.jvs.2010.05.019. Epub 2010 Jul 13. PMID 20630688
- [Background] Sevestre MA, Quashie C, Genty C, Rolland C, Quere I, Bosson JL; Optimev study investigators. Clinical presentation and mortality in pulmonary embolism: the Optimev study. J Mal Vasc. 2010 Jul;35(4):242-9. doi: 10.1016/j.jmv.2010.05.004. Epub 2010 Jul 2. PMID 20598461
- [Background] Sevestre MA, Labarere J, Casez P, Bressollette L, Haddouche M, Pernod G, Quere I, Bosson JL. Outcomes for inpatients with normal findings on whole-leg ultrasonography: a prospective study. Am J Med. 2010 Feb;123(2):158-65. doi: 10.1016/j.amjmed.2009.05.034. PMID 20103025
- [Background] Casez P, Labarere J, Sevestre MA, Haddouche M, Courtois X, Mercier S, Lewandowski E, Fauconnier J, Francois P, Bosson JL. ICD-10 hospital discharge diagnosis codes were sensitive for identifying pulmonary embolism but not deep vein thrombosis. J Clin Epidemiol. 2010 Jul;63(7):790-7. doi: 10.1016/j.jclinepi.2009.09.002. Epub 2009 Dec 2. PMID 19959332
- [Background] Galanaud JP, Sevestre-Pietri MA, Bosson JL, Laroche JP, Righini M, Brisot D, Boge G, van Kien AK, Gattolliat O, Bettarel-Binon C, Gris JC, Genty C, Quere I; OPTIMEV-SFMV Investigators. Comparative study on risk factors and early outcome of symptomatic distal versus proximal deep vein thrombosis: results from the OPTIMEV study. Thromb Haemost. 2009 Sep;102(3):493-500. doi: 10.1160/TH09-01-0053. PMID 19718469
- [Background] Sevestre MA, Labarere J, Casez P, Bressollette L, Taiar M, Pernod G, Quere I, Bosson JL. Accuracy of complete compression ultrasound in ruling out suspected deep venous thrombosis in the ambulatory setting. A prospective cohort study. Thromb Haemost. 2009 Jul;102(1):166-72. doi: 10.1160/TH09-01-0048. PMID 19572082
- [Background] Constans J, Salmi LR, Sevestre-Pietri MA, Perusat S, Nguon M, Degeilh M, Labarere J, Gattolliat O, Boulon C, Laroche JP, Le Roux P, Pichot O, Quere I, Conri C, Bosson JL. A clinical prediction score for upper extremity deep venous thrombosis. Thromb Haemost. 2008 Jan;99(1):202-7. doi: 10.1160/TH07-08-0485. PMID 18217155
- [Background] Sevestre MA, Labarere J, Brin S, Carpentier P, Constans J, Degeilh M, Deslandes B, Elgrishi I, Lanoye P, Laroche JP, Le Roux P, Pichot O, Quere I, Bosson JL; OPTIMEV study. [Optimizing history taking for evaluating the risk of venous thromboembolism: the OPTIMEV study]. J Mal Vasc. 2005 Sep;30(4 Pt 1):217-27. doi: 10.1016/s0398-0499(05)88206-x. French. PMID 16292199